CLINICAL TRIAL: NCT03097575
Title: Bronchial NIR Image-guided Resection, Mapping And Targeted Lymphadenectomy for Lung Lesions
Brief Title: Bronchial NIR Image-guided Resection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Society of University Surgeons (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Yolonda Colson, MD, PhD, Dr., Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014P001436
Record Dates: First submitted 2017-03-13; First posted 2017-03-31 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Sentinel Lymph Node
Keywords: Lung lesions; Navigational bronchoscopy; Near infrared imaging; Lymphadenectomy
MeSH Terms: interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ICG Intervention (Experimental): The intervention to be administered is the indocyanine green for NIR Lymphatic Mapping. All study subjects will receive this same intervention; there is only one arm.
  Interventions: Drug: ICG Intervention; Device: Near Infrared Imaging

INTERVENTIONS:
Drug: ICG Intervention — Patients enrolled in the study will undergo injection of near infrared dye indocyanine green around the lung lesion or within the adjacent segmental bronchus at the time of surgery via navigational bronchoscopy, or if not amenable to navigational bronchoscopy injection, then injection will be carried out via a transthoracic approach through the incision or under CT-guidance.
  Other Names: NIR Lymphatic Mapping; Indocyanine Green
Device: Near Infrared Imaging — A near-infrared camera device will be used to detect indocyanine green following injection.

SUMMARY:
This is a clinical trial to evaluate the use of peritumoral injection of near-infrared dye indocyanine green to identify lung lesions and sentinel lymph nodes. The primary purpose is to determine if the use of ICG injected via navigational bronchoscopy, CT-guided or transthoracic allows us to identify the first lymph node that drains from the tumor, and thus would be the most likely site for metastatic disease, and remove it for analysis to improve the ability to detect tumor in this node and to remove this additional site that potentially contains tumor cells. Using this intraoperative imaging technique, we aim to improve the identification of lung nodules for resection and the intraoperative identification of sentinel lymph nodes in the event that a lymphadenectomy is performed.

DETAILED DESCRIPTION:
Patients enrolled in the study will undergo peritumoral injection of near-infrared dye indocyanine green around the lung lesion or within the adjacent segmental bronchus at the time of surgery. ICG injection will be carried out via navigational bronchoscopy, CT-guided or trans-thoracic ICG injection (dependent on lesion location) and ICG imaging of the sentinel lymph nodes will be undertaken using an NIR-enabled camera.

* This study is designed primarily to determine the safety and feasibility of intra-operative localization of thoracic lesions following ICG injection, and second, to include an assessment of the predictive value of sentinel lymph nodes relative to the disease status of the greater lymphadenectomy specimen as well as disease recurrence rates.
* We are using a dose approximately 100 times lower than previously approved for injection in the blood. After a few minutes, the surgeon will look at these lymph nodes with near-infrared fluorescence and then remove any fluorescent and non-fluorescent lymph nodes near the tumor, as is standard for lung surgery.
* The "filtered" near-infrared light causes the indocyanine green dye to fluoresce so that the surgeon can identify the lymph nodes most likely to contain tumor cells. If the lymph node is not found in the group of nodes usually removed, we will use the near-infrared light to look near the tumor for the sentinel lymph nodes and guide the surgeon so that the sentinel nodes can be removed and studied. The surgeon will then continue with the operation and remove the tumor. The lymph nodes are processed for special analysis tailored to finding metastasis in sentinel lymph nodes.
* As is standard of care, patients will be monitored for evidence of recurrence by their surgeon. Recurrences will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have agreed to undergo video assisted thoracoscopic surgery or thoracotomy for surgical resection as recommended by their thoracic surgeon.
* 18 years of age or older
* Documented, signed, dated informed consent obtained prior to any study specific procedures being performed

Exclusion Criteria:

* Pregnant women are excluded and women of childbearing potential without a negative pregnancy test prior to study procedures. All patients with Iodine allergies will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01-06 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (safety and feasibility) of intraoperative NIR-image-guided localization of lung lesions using peritumoral ICG injection. | 5 years
  In this initial proof-of-concept pilot trial for patients undergoing surgical resection of a suspicious lung lesion, we will translate the new technology of NIR-imaging to the OR and assess safety and feasibility of ICG delivery, optimize the ability to "NIR tattoo" and visualize lung lesions for targeted resection vs NIR-highlighted segmental resections, assess histology of the surgical margin and determine lesional characteristics which predict successful NIR imaging. Safety and feasibility will be measured quantitatively by the number of participants with treatment-related adverse events, as assessed by CTCAE v4.0.

SECONDARY OUTCOMES:
Investigate whether SLNs can be identified using NIR-guidance following peritumoral ICG injection. | 5 years
  Technical difficulty and clinical complications have resulted in < 50% of surgeons performing complete removal of tumor draining lymph nodes at the time of surgery. Therefore, we will assess the feasibility of SLN identification following ICG injection for "targeted" lymph node sampling and focused analysis staging. This Outcome will be addressed only in cases where a lymphadenectomy is performed.
Assess if NIR image-guided SLN excision enhances detection of metastatic disease and whether the presence of untreated occult metastatic disease/mutational analysis of primary tumors/secondary sites of disease including SLNs are predictors of outcome | 5 years
  Studies in stage I and II lung cancer have demonstrated "occult" nodal metastatic disease affects clinical outcomes, however, currently there is no accurate means to identify micrometastatic nodal disease in these patients prospectively. Therefore, we will analyze the SLN results to determine whether prospectively identified "occult" micrometastatic disease in the SLN is a "predictor" of disease recurrence. This Outcome is pertinent only to cases in which a lymphadenectomy was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Yolonda L Colson, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers at this time.